CLINICAL TRIAL: NCT04212143
Title: Central Blood Pressure and Pulse Wave Velocity in Children With and Without Kidney Transplants
Brief Title: Central Blood Pressure and Pulse Wave Velocity in Kidney Transplant Recipients
Status: Active, not recruiting | Type: Observational
Sponsor: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Kristen Sgambat, Clinical Dietitian IV, Children's National Research Institute
Other Study IDs: Pro00013491
Record Dates: First submitted 2019-12-23; First posted 2019-12-26 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- children with kidney disease: Kidney transplant recipients age 3 to 21 years
  Interventions: Other: there is no intervention
- healthy control: Healthy children age 3 to 21 years
  Interventions: Other: there is no intervention

INTERVENTIONS:
Other: there is no intervention — There is no intervention in this study. It is observational only.

SUMMARY:
An observational cohort study will be conducted to non-invasively investigate central blood pressure and pulse wave velocity in children with kidney disease and controls. Using an oscillometric monitor, the investigators aim to non-invasively obtain the central blood pressure and pulse wave velocity (PWV), or arterial stiffness, of children with kidney disease. The investigators will also enroll age- and race-matched healthy controls and measure the same parameters for comparison. In addition, the investigators will measure PWV by standard arterial tonometry method in a subset of patients.

DETAILED DESCRIPTION:
The specific aims of the study are as follows:

1. Using an oscillometric blood pressure monitor, the investigators aim to non-invasively obtain the central blood pressure and pulse wave velocity (PWV), or arterial stiffness, of children with kidney disease.
2. Measure oscillometric central blood pressure and PWV in age and race matched healthy children.
3. Measure PWV by standard arterial tonometry method in a subset of patients, and compare these measurements to the PWV measured using the oscillometric device.
4. Measure body composition of patients and controls (Body Mass Index, Waist-to-Height ratio, %body fat, and mid-arm muscle circumference) to see how this relates to central blood pressure and PWV.

ELIGIBILITY:
Inclusion Criteria:

* kidney transplant recipients who are at least 6 months post-transplant
* healthy children matched for age sex and race

Exclusion Criteria:

* age less than 3 years

Ages: 3 Years to 21 Years | Sex: All
Age Groups: Child, Adult
Study Population: pediatric kidney transplant recipients and healthy controls
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Oscillometric central blood pressure | cross-sectional measurement performed in patients who are between 6 months to 10 years post-transplant
  Central blood pressure as measured by oscillometric blood pressure device
Oscillometric pulse wave velocity | cross-sectional measurement performed in patients who are anywhere between 6 months to 10 years post-transplant
  Pulse wave velocity as measured by oscillometric blood pressure device

SECONDARY OUTCOMES:
Body mass index (BMI) in kg/m2 | cross-sectional measurement performed in patients who are anywhere between 6 months to 10 years post-transplant
  weight measured in kg and height measured in cm will be combined to determine BMI (kg/m2)
Waist circumference (cm) | cross-sectional measurement performed in patients who are anywhere between 6 months to 10 years post-transplant
  waist circumference will be measured in cm using a flexible tape measure
Mid arm circumference (cm) | cross-sectional measurement performed in patients who are anywhere between 6 months to 10 years post-transplant
  Mid arm circumference will be measured in cm using a flexible tape measure

CONTACTS AND LOCATIONS:
Locations (1):
- Children's National Medical Cetner, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No